CLINICAL TRIAL: NCT04045717
Title: Hypofractionated Focal Lesion Ablative Microboost in prostatE Cancer 2.0
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: The Netherlands Cancer Institute (Other); Radboud University Medical Center (Other); Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S63033
Record Dates: First submitted 2019-07-19; First posted 2019-08-05 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Prostate Adenocarcinoma; Prostate Cancer; Prostate Neoplasm
Keywords: Stereotactic Body Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypo-FLAME 2.0 (Experimental): SBRT technique with 35 Gy in 5 fractions to the whole prostate gland and an additional simultaneously integrated focal boost to the tumor nodule(s) visible on MRI up to 50 Gy (overall treatment time (OTT) = 15 days).
  Interventions: Radiation: Hypo-FLAME 2.0 study

INTERVENTIONS:
Radiation: Hypo-FLAME 2.0 study — SBRT technique with 35 Gy in 5 fractions to the whole prostate gland and an additional simultaneously integrated focal boost to the tumor nodule(s) visible on MRI up to 50 Gy (overall treatment time (OTT) = 15 days).

SUMMARY:
The hypo-FLAME 2.0 study is a multicenter phase II study (n=124) investigating the feasibility and safety of a reduction in the overall treatment time of radiotherapy for prostate cancer patients, making use of hypofractionated stereotactic body radiotherapy with focal boosting. We are looking for the optimal overall treatment time for this treatment strategy in the Hypo-FLAME 2.0 trial. In this study the total treatment time will be halved (15 days) in comparison with the total treatment time in the former hypo-FLAME trial (29 days) (NCT02853110).

DETAILED DESCRIPTION:
Rationale: External beam radiotherapy is one of the standard treatment options for patients with prostate cancer. The overall treatment time of a standard fractionated schedule varies between 7 and 8 weeks (i.e. 35-40 fractions, 5x/week). Recent studies have identified a proportionally longer overall treatment time as a potential adverse factor for treatment outcome in prostate cancer patients who were treated by conventional radiotherapy schedules. Furthermore shortening of the overall treatment time promotes patient convenience. An extreme shortening of the overall treatment time is possible by using hypofractionated treatment schedules with simultaneous integrated intraprostatic tumor boosting to overcome local recurrences.

Objective: In this study we will investigate the feasibility and safety of a reduction in the overall treatment time of radiotherapy for prostate cancer patients, making use of hypofractionated stereotactic body radiotherapy with focal boosting. We are looking for the optimal overall treatment time for this treatment strategy in the Hypo-FLAME 2.0 trial. In this study the total treatment time will be halved (15 days) in comparison with the total treatment time in the former Hypo-FLAME trial (29 days). Besides a potential biological advantage, the reduced overall treatment time offers benefits with respect to patient convenience.

Study population: One hundred twenty four patients with histologically proven intermediate- or high-risk prostate cancer will be included in this multicenter phase II study. Patients referred for external beam radiotherapy who fulfil the inclusion criteria and without any of the exclusion criteria will be included in the present trial after written informed consent.

Intervention: Patients will be treated with a stereotactic body radiation therapy technique up to 35 Gray in 5 fractions of 7 Gray to the whole prostate gland. Additionally a simultaneously integrated focal boost to the macroscopic tumor nodule(s) visible on MRI up to 50 Gray (10 Gray/fraction) will be delivered. Treatment fractions will be delivered twice weekly, resulting in an overall treatment time of 2,5 weeks.

Main study endpoints: The primary endpoint of this study is acute gastrointestinal and genitourinary toxicity, scored using the Common Terminology Criteria Adverse Events version 5.0. Secondary endpoints are late gastrointestinal and genitourinary toxicity, quality of life and biochemical disease free survival defined by the Phoenix consensus definition.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 18 years with histologically confirmed prostate adenocarcinoma
* Intermediate- or high-risk PCa, defined as at least one of the following risk criteria:

  * Clinical stage: T2b, T2c, T3a or T3b with less than 5 mm invasion in the seminal vesicles (defined on MRI) N0 M0
  * Gleason sum score ≥ 7
  * PSA ≥ 10 ng/mL.
* Prostate tumor nodule visible on mpMRI
* Ability to give written informed consent and willingness to return for follow-up

Exclusion Criteria:

* Prior pelvic radiotherapy or transurethral prostate resection
* Unsafe to have gold fiducial marker implantation, if gold fiducial markers are used for image guidance (non MR-linac)
* Contraindications to MRI according to the Radiology Department guidelines (metal implants, non-compatible cardiac device, allergy to gadolinium, severe renal dysfunction or severe claustrophobia)
* World Health Organization (WHO) performance score > 2
* International prostate symptoms score (IPSS score) ≥ 15
* PSA > 30 ng/mL

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2032-02-16 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 90 days after first radiation treatment
  Acute toxicity is scored using the Common Terminology Criteria Adverse Events version 5.0.

SECONDARY OUTCOMES:
Late toxicity | 10 years after first radiation treatment
  Late toxicity is scored using the Common Terminology Criteria Adverse Events version 5.0.
Quality of life - general | 5 years after first radiation treatment
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire
Quality of life - prostate specific | 5 years after first radiation treatment
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-PR25 questionnaire
Biochemical disease free survival | 10 years after first radiation treatment
  Biochemical disease free survival is defined by the Phoenix consensus definition.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Haustermans, M.D. PhD, Principal Investigator — UZ Leuven
Locations (3):
- University Hospitals Leuven, Leuven, Belgium
- Netherlands (2):
  - The Netherlands Cancer Institute, Amsterdam
  - Radboudumc, Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] De Cock L, Draulans C, Pos FJ, Isebaert S, De Roover R, van der Heide UA, Smeenk RJ, Kunze-Busch M, van der Voort van Zyp J, de Boer H, Kerkmeijer LGW, Haustermans K. From once-weekly to semi-weekly whole prostate gland stereotactic radiotherapy with focal boosting: Primary endpoint analysis of the multicenter phase II hypo-FLAME 2.0 trial. Radiother Oncol. 2023 Aug;185:109713. doi: 10.1016/j.radonc.2023.109713. Epub 2023 May 11. PMID 37178932